CLINICAL TRIAL: NCT00691626
Title: CBT for Nightmares in OEF/OIF Veterans
Brief Title: Cognitive Behavioral Therapy (CBT) for Nightmares in Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT074364
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Posttraumatic Stress Disorder; Sleep Disorders; Nightmares
Keywords: posttraumatic stress; nightmares; sleep; psychotherapy; imagery rehearsal; insomnia; behavioral treatment; veterans; Operation Iraqi Freedom; Operation Enduring Freedom
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial comparing two forms of psychotherapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: CBT for Insomnia plus Imagery Rehearsal (Experimental): CBT for Insomnia plus Imagery Rehearsal
  Interventions: Behavioral: CBT for Insomnia plus Imagery Rehearsal
- Arm 2: CBT for Insomnia (Active Comparator): CBT for Insomnia
  Interventions: Behavioral: CBT for Insomnia plus psychoeducation

INTERVENTIONS:
Behavioral: CBT for Insomnia plus Imagery Rehearsal — patients receive standard CBT for insomnia and psychoeducation combined with techniques of imagery rehearsal aimed at reducing posttraumatic nightmare frequency and distress
  Arms: Arm 1: CBT for Insomnia plus Imagery Rehearsal
Behavioral: CBT for Insomnia plus psychoeducation — patients receive standard CBT for insomnia combined with psychoeducation
  Other Names: Sleep and Nightmare Management
  Arms: Arm 2: CBT for Insomnia

SUMMARY:
The purpose of this study is to compare the effectiveness of two talk therapies for OEF/OIF Veterans at the Michael J. Crescenz and the West Haven VA Medical Centers. Participants will randomly receive one of two individual treatments intended to improve the sleep disturbance and nightmares of returning Veterans.

DETAILED DESCRIPTION:
This is a dismantling study with the objective of determining whether imagery rehearsal is essential to the efficacy of imagery rehearsal + CBT-I for improving the sleep and nightmare disturbance in Veterans with PTSD and recurrent nightmares.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in treatment in the Michael J. Crescenz VA Medical Center or VA Connecticut Healthcare System Mental Health Clinic
* Meets DSM-IV-R criteria for current PTSD (within the past month)
* Repetitive, military-related nightmares (at least 1 every 2 weeks, for at least 6 months)
* A global sleep disturbance, as indicated by a score of five or greater on the Pittsburgh Sleep Quality Index
* Ability to read and speak English
* A concurrent anxiety disorder or depressive disorder diagnosis will be allowed
* Dementia related to head injury and amnestic disorder related to head injury will be allowed

Exclusion Criteria:

* Current substance dependence
* Bipolar disorder
* Delirium
* Dementia that is not related to head injury
* Amnestic disorder that is not related to head injury
* Schizophrenia and other psychotic disorders
* Severe traumatic brain injury, as indicated by self-report (loss of consciousness or alteration of mental status greater than 24 hours, or peri-traumatic memory loss, or any posttraumatic amnesia greater than 7 days)
* The presence of diagnosed sleep disorders other than insomnia: narcolepsy, circadian rhythm sleep disorders, and periodic limb movement disorder. Participants in treatment for sleep apnea, or who have not benefited from or declined available treatment may be included.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Nightmare Frequency Questionnaire, Nightmare Distress Questionnaire | post-treatment, 3 month and 6-month follow-up
  The NFQ measures the number of nightmares/week and the number of nights with a nightmare/week.
  The NDQ measures the distress associated with nightmare experiences.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | post-treatment, 3 month and 6-month follow-up
  This is a standard instrument for measuring basic sleep parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Ross, MD PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA; Ilan Harpaz-Rotem, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scott JC, Harb G, Brownlow JA, Greene J, Gur RC, Ross RJ. Verbal memory functioning moderates psychotherapy treatment response for PTSD-Related nightmares. Behav Res Ther. 2017 Apr;91:24-32. doi: 10.1016/j.brat.2017.01.004. Epub 2017 Jan 13. PMID 28110112
- [Result] Harb GC, Cook JM, Phelps AJ, Gehrman PR, Forbes D, Localio R, Harpaz-Rotem I, Gur RC, Ross RJ. Randomized Controlled Trial of Imagery Rehearsal for Posttraumatic Nightmares in Combat Veterans. J Clin Sleep Med. 2019 May 15;15(5):757-767. doi: 10.5664/jcsm.7770. PMID 31053215